CLINICAL TRIAL: NCT03381677
Title: A Prospective, Multi-Center, Randomized Concurrently Controlled Trial to Evaluate the Safety and Effectiveness of the Altum® Pedicle Osteotomy System for Use in Lumbar Spinal Stenosis
Brief Title: Pedicle Osteotomy for Stenosis Trial
Acronym: POST
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: In light of the ongoing COVID-19 pandemic and its impact on clinical trials
Sponsor: Innovative Surgical Designs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-2016-01
Record Dates: First submitted 2017-11-28; First posted 2017-12-22 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Lumbar Spinal Stenosis; Spondylolisthesis, Grade 1; Neurogenic Claudication
Keywords: pedicle lengthening osteotomy; spinal stenosis; decompression
MeSH Terms: conditions — Spinal Stenosis; Spondylolisthesis; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Pedicle Lengthening Osteotomy (Experimental): Lumbar decompressive surgery via Pedicle Lengthening Osteotomy Procedure with the Altum® Device
  Interventions: Device: Pedicle Lengthening Osteotomy with Altum® Device
- Control group (Active Comparator): Decompressive surgery via open surgical decompression and Transforaminal Lumbar Interbody Fusion (TLIF) using either a midline or paramedian incision with implantation of bilateral pedicle screws (4 screws) and rods (2 rods) and an interbody fusion cage (1 PEEK fusion cage, coated or uncoated):
  1. DePuy Synthes Expedium® 5.5 System, Stryker Xia 5.5 System, Medtronic CD Horizon Solera 5.5 Systemor Innovative Surgical Designs True Spinal Fixation System; and
  2. DePuy Synthes Concord TLIF cage, Stryker UniLIF TLIF cage, Medtronic Capstone TLIF cage or Meditech Talos TLIF cage.
  Interventions: Device: Control

INTERVENTIONS:
Device: Pedicle Lengthening Osteotomy with Altum® Device — Decompressive surgery via Pedicle lengthening osteotomy using Altum Device. Altum is intended for pedicle lengthening to correct degenerative lumbar spinal stenosis in the presence of a grade 1 degenerative spondylolisthesis. The Altum bone saw is designed for creating an osteotomy at the base of each pedicle. The Altum implant is designed for distraction of the pedicle osteotomy and for lengthening of the pedicles. Altum is appropriate for skeletally mature adults with symptomatic stenosis at one or two levels between L2-L5.
  Arms: Pedicle Lengthening Osteotomy
Device: Control — Decompressive surgery via open surgical decompression and Transforaminal Lumbar Interbody Fusion (TLIF) using either a midline or paramedian incision with implantation of bilateral pedicle screws (4 screws) and rods (2 rods) and an interbody fusion cage (1 PEEK fusion cage, coated or uncoated):
  1. DePuy Synthes Expedium® 5.5 System, Stryker Xia 5.5 System, Medtronic CD Horizon Solera 5.5 Systemor Innovative Surgical Designs True Spinal Fixation System; and
  2. DePuy Synthes Concord TLIF cage, Stryker UniLIF TLIF cage, Medtronic Capstone TLIF cage or Meditech Talos TLIF cage.
  Arms: Control group

SUMMARY:
This is a pivotal Randomized Clinical trial to compare the safety and effectiveness of the Pedicle Lengthening Osteotomy Procedure with implantation of the Altum® Device to open surgical decompression and Transforaminal Lumbar Interbody Fusion (TLIF) in patients with symptomatic, one or two level lumbar spinal stenosis (LSS) and one level grade I degenerative spondylolisthesis requiring surgical treatment.

DETAILED DESCRIPTION:
LSS is a narrowing of the spinal canal and/or the intervertebral foramina by bony spurs or soft tissues that decrease space for the neural elements resulting in compression of the nerve roots or spinal cord in the lumbar region of the spine. LSS can cause low back pain, weakness, numbness, and pain and loss of sensation in the buttocks and legs. In most cases the symptoms improve when the patient is sitting or leaning forward, due to the flexed position of the vertebra which leads to reduced impingement of the neural tissue. In addition, many patients with LSS complain of pain when standing and walking referred to as neurogenic intermittent claudication (NIC). Nonsurgical management is well-established as the first-line treatment approach for LSS patients with mild to moderate symptoms. It typically involves the prescription of modified physical activity, physiotherapy, anti-inflammatory drugs, epidural steroid injections, use of a lumbar corset or some combination thereof.

Surgical treatment is reserved for patients who do not obtain adequate relief of symptoms by conservative management. The goal of surgical treatment for LSS is to relieve the compression of the spinal nerves in the spinal canal or neural foramina. Such decompressive surgery generally involves laminectomy, laminotomy, foraminotomy, partial facetectomy or some combination thereof. Decompressive surgery in subjects with LSS and spondylolisthesis commonly requires fusion to stabilize the spondylolisthesis. The most commonly performed lumbar fusion for patient's with the combination of LSS and spondylolisthesis is a Transforaminal Lumbar Interbody Fusion (TLIF) which involves stabilizing the motion segment by placing pedicle screws, rods and an interbody fusion cage. Autograft or allograft bone are commonly used to bring about fusion or a bridging of bone across the intervertebral joint.

The Altum® Pedicle Osteotomy System contains the implants and instruments required to perform the pedicle lengthening osteotomy procedure for the treatment of LSS. The Altum® implant is an expandable bone screw that is available in a variety of sizes (7.5 mm, 8.5 mm and 9.5 mm). Altum® instruments are manufactured from IXEF PARA GS-1022 GY/51, medical grade titanium alloy (Ti 6AL-4V ELI ASTM F-136), and medical grade stainless steel (17-4 ASTM F899).

ELIGIBILITY:
Inclusion Criteria:

1. Is a male or female patient between 40 and 80 years of age.
2. Has the diagnosis of degenerative spinal stenosis of the lumbar region (defined as L2-L5), defined by one or more of the following: a) narrowingof the mid-sagittal spinal canal (central stenosis), b) narrowing between the facet superior articular process (SAP) and the posterior intervertebral disc margin (lateral recess stenosis), c) narrowing of the nerve root foraminal canal(s) (foraminal stenosis) and has, at the same level, radiographic confirmation on plain lateral flexion/extension radiographs of a degenerative grade I spondylolisthesis at the same level, defined as at least 1% but not greater than 25%, offset between the posterior margins of the adjacent vertebral bodies at the index level.
3. Neurogenic claudication or radiculopathic symptoms including leg pain, muscle weakness, and/or sensation abnormality, with or without back pain, which is worse with extended posture and relieved by flexion, as evidenced by patient history.
4. Has pain in the leg and/or buttock that is worse with standing as compared to sitting.
5. Has radiographic confirmation on CT or MRI of moderate or greater lumbar spinal stenosis at the index level defined as > 25% reduction in area of the central and/or lateral recess and/or foraminal regions of the spinal canal as compared to the adjacent level.
6. Has radiographic confirmation on CT or MRI of compression of the thecal sac and/or cauda equina and/or nerve root(s) due to hypertrophy of the facet joints and/or ligamentum flavum thickening/buckling
7. Has undergone a 6 month or longer course of conservative therapy without sufficient relief of symptoms that has included one or more of the following interventions: physical therapy, bracing, systemic and/or injected medications.
8. Has moderate or greater impairment on the Zurich Claudication Questionnaire (ZCQ) Physical Function scale (PF) defined as a score of 2 or greater.
9. Has moderate or greater impairment on the Oswestry Disability Index defined as a score of 30 or greater.
10. Is a surgical candidate for lumbar decompressive surgery at one or two levels in the L2 through L5 region of the spine.
11. Is psychosocially, mentally and physically able to comply with all study procedures required by the study protocol including attending all scheduled visits and interventions.
12. Is able to provide voluntary, informed consent to participate in the clinical trial and has signed the informed consent documents.

Exclusion Criteria:

1. Has had prior spinal surgery at any level between L1 and S1.
2. Requires more than 2 lumbar levels of surgical decompression.
3. Has a degenerative spondylolisthesis of greater than grade I defined as greater than 25% offset between the posterior margins of adjacent vertebral bodies on plain lateral flexion/extension radiographs or does not have a grade I degenerative spondylolisthesis, defined as 0% offset between the posterior margins of adjacent vertebral bodies on a plain lateral flexion/extension radiograph.
4. Has more than one level of degenerative spondylolisthesis or has spondylolisthesis located at lumbar levels which are not treated with surgical decompression. Has the diagnosis of peripheral neuropathy.
5. Has a complete motor or sensory deficit.
6. Has a pars defect.
7. Has facet joints at the implant level that are absent or fractured.
8. Has lumbar scoliosis with a Cobb angle of greater than 25o.
9. Has a disc herniation at any lumbar level requiring surgical intervention.
10. Has symptomatic hip arthritis or hip pain.
11. Has a Body Mass Index (BMI) of greater than 40.
12. Has a known allergy to titanium or titanium alloys.
13. Has osteoporosis. The SCORE (Simple Calculated Osteoporosis Risk Estimation) will be used to screen subjects who require DEXA; Subjects with T-score < -2.5 (per The World Health Organization definition) will be excluded.
14. Has a history of Paget's disease, osteomalacia, or any other metabolic bone disease.
15. Has a history of rheumatoid arthritis or other systemic autoimmune disease.
16. Requires medications or drugs known to interfere with bone/soft tissue healing (e.g., chronic systemic corticosteroids). Corticosteroids used for 6 weeks or less are not an exclusion criteria.
17. Has insulin dependent diabetes mellitus.
18. Has cauda equina syndrome, defined as neural compression in the lumbar spine causing neurogenic bowel (rectal incontinence) or neurogenic bladder (bladder retention or incontinence) dysfunction.
19. Only has axial back pain with no leg or buttock pain.
20. Has back or leg pain of unknown etiology.
21. Has evidence or the diagnosis of significant peripheral vascular disease (e.g. diminished or absent dorsalis pedis or posterior tibial pulses)
22. The patient currently has any of the following: schizophrenia, bipolar disorder, major depression, major psychotic disorder, and substance or alcohol abuse or dependency as defined by the DSM V.
23. Has participated in a clinical trial of another investigational drug or device within the past 2 years.
24. Has an active, chronic infection, either systemic or local.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2017-10-26 (Actual); Primary Completion 2022-10-26 (Estimated); Study Completion 2024-10-26 (Estimated)

PRIMARY OUTCOMES:
Zurich Claudication Questionnaire (ZCQ) | 24 months
  Clinically significant improvement in outcomes ZCQ scores compared to baseline
  * Improvement in physical function by > 0.5 points
  * Improvement in symptom severity by > 0.5 points
  * "Satisfied" or "somewhat satisfied" as defined by a score of < 2.5 points on the patient satisfaction domain
No reoperations | Index level
  No re-operations, removals, revisions or supplemental fixation at the index level.
Adjacent level surgery | 24 months
  No additional surgery at the adjacent levels
Adverse events | 24 months
  No major device-related adverse events
Radiological Success | 24 months
  Presence of continuous bridging bone across both pedicle osteotomy sites on CT scanning,
  * No evidence of bridging bone between the upper and lower vertebral endplates on CT scanning, and evidence of continued motion as demonstrated on flexion-extension films
  * Absence of a major device related adverse event (device breakage, disassembly or migration)

SECONDARY OUTCOMES:
Oswestry Disability Index | 24 months
  Improvement in Oswestry Disability Index v2.1a > 15 points from baseline to 24 months
EQ5D | 24 months
  Change in EQ5D from baseline to 24 months
SF-12 | 24 months
  Change in SF-12v2.0™ from baseline to 24 months
Pain Visual Analog Scale (VAS) for Back and Leg | 24 months
  Pain Visual Analog Scale (VAS) is a measure of pain intensity. It is a continuous scale comprised of a 100mm line ranging from 0 (no pain) to 10 (worst imaginable pain). Patients mark a line on the scale depicting their pain level. A VAS score is determined by measuring where the mark is made relative to the ends of the line. VAS will be done separately for low back, right leg and left leg pain.Improvement in VAS for back, right leg and left leg pain of 20/100mm from baseline to 24 months
Cost | Index surgery
  Direct costs of the episode of care
Opioid use | baseline to 24 months
  Use of opioid analgesics
Return to work | Anytime from discharge after surgery up to 24 months (+/- 60 days)
  Patient will report the date of which they return to work
Daily activities | baseline to 24 months
  Time for return to usual daily activities
Patient Satisfaction | 24 months
  A series of questions intended to assess the effects of the procedure itself on your well-being, and does not refer to the hospital or its staff. One out of 5 statements will be chosen based on the patient's level of satisfaction: The procedure results met my expectations and I feel better than I did before surgery; The procedure improved my condition enough that I would go through it again for the same outcome; The procedure helped me but I would not go through it again for the same outcome; I feel the same or worse compared to before surgery.
  Furthermore, patients will be ask to choose one statement based on how they feel today compared to their last visit: I feel much better; I feel somewhat better; I feel somewhat worse; I feel much worse.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Rinehart, Study Director — Sponsor GmbH
Locations (1):
- Rothman Institute, Bryn Mawr, Pennsylvania, United States